CLINICAL TRIAL: NCT05155462
Title: Analysis of the Different Strategies for Revascularization of the Lower Limbs by Peripheral Angioplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A00868-47
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Peripheral Arterial Disease; Angioplasty
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient treated for defined symptomatic chronic lower extremity ischemia
  Interventions: Other: One or two phone call

INTERVENTIONS:
Other: One or two phone call — Phone call to collect patient data

SUMMARY:
Peripheral arterial disease (PAD) caused by atherosclerosis causes damage to the arteries originating in the aorta (descending) from the iliacs to the extremities of the lower limbs. It causes significant morbidity and mortality. Percutaneous revascularization plays a key role in the management of these patients. Many percutaneous treatment options have been developed: arteriectomy, naked stents, active balloons and active stents. Of these, only paclitaxel-active stents were successful in reducing the rates of restenosis and reoperation in patients with superficial femoral artery injury.The main objective is to study symptomatic improvement at 1 year of patients treated with revascularization of the lower limbs.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated by the peripheral angioplasty department of Claude Galien Hospital from January 2010 and with at least 1 year of follow-up after the revascularization procedure
* Patient treated for symptomatic chronic ischemia of the lower limbs defined by Rutherford categories 2-4 and / or Leriche stage greater than 2a
* Stenosis or restenosis (history of balloon angioplasty, active balloon or bare stent)
* Degree of stenosis ≥ 50% by angiographic evaluation visual, by CT scan or by Doppler ultrasound
* Patient affiliated or beneficiary of a social security scheme
* Patient aged 18 or over
* Patient having been informed and not opposing this research

Exclusion Criteria:

* Medical history of myocardial infarction or stroke within 3 months of the revascularization procedure
* Unstable angina at the time of the revascularization procedure
* Sepsis at the time of the revascularization procedure
* Major under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Hospitalized without consent
* Pregnant, breastfeeding or parturient woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient 18 or over, treated for symptomatic chronic ischemia of the lower limbs defined by Rutherford categories 2-4 and / or Leriche stage greater than 2a
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2021-12-09 (Estimated)

PRIMARY OUTCOMES:
Symptomatic improvement will be assessed by the evolution of the Leriche and Rutherford classifications before the revascularization procedure and 1 year after the revascularization procedure | 1 year
  Lerich classification : stage I to IV Rutherford : stage 0 to 6

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Claude Galien, Quincy-sous-Sénart, France